CLINICAL TRIAL: NCT03964987
Title: PDX-1 and NGN-3 Expression in Gestational Diabetes
Brief Title: Pancreatic Duodenal Homeobox Factor-1 (PDX-1) and Neurogenin-3 (NGN-3) in Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: 2016-09-481
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Gestational Diabetes
Keywords: PDX-1; NGN-3; Glucose
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Women with normoevolutionary gestation.
- Problem group: Patients with GDM.

SUMMARY:
Introduction: Depletion of the ability of the cells ß to secrete the amount of insulin required by pregnancy, increasing the risk of develop Gestational Diabetes Mellitus (GDM). The aim was to contrast the messenger RNA (mRNA) expression of the pancreatic duodenal homeobox factor-1 (PDX-1) and Neurogenin-3 (Ngn-3) in peripheral blood of pregnant women with GDM versus women with normal pregnancies.

Material and methods: This was a prospective, clinical and cross-sectional study, conforming two groups of pregnant women: a) patients with a healthy gestation and b) patients with GDM. Besides anthropometry and routine laboratorial test, real-time polymerase chain reaction (Real-Time PCR), was used to quantify the expression of PDX-1 and NGN-3.

DETAILED DESCRIPTION:
Pregnant women attended in the Maternal-Fetal Medicine Service of the "Mónica Pretelini Sáenz" Maternal-Perinatal Hospital, were invited to participate. Those with autoimmune diseases, heart disease, nephropathy, liver disease or any other chronic condition were excluded and those with incomplete clinical files were discarded from the final analysis. Two groups were integrated: a) patients with a healthy gestation and b) patients with GDM.

From all patients the next information was captured in an excell sheet: weight, height, Body Mass Index, blood pressure, albumin, creatinine, electrolytes, glucose, total cholesterol, triglycerides, transaminases and relative expression of PDX-1 and NGN-3.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women older than 18 years old.

Exclusion Criteria:

* Those with autoimmune diseases, heart disease, nephropathy, liver disease or any other chronic condition.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women attended in the Maternal-Fetal Medicine Service of the HMPMP.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ARNm expression | Nine months
  Expression of the genes PDX-1 and NGN-3

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Principal Investigator — Maternal-Perinatal Hospital "Mónica Pretelini Sáenz"
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Information will be available upon request.

REFERENCES:
- [Background] Sandikci M, Karagenc L, Yildiz M. Changes on the Pancreas in Experimental Diabetes and the Effect of Lycopene on These Changes: Pdx-1, Ngn-3, and Nestin Expressions. Anat Rec (Hoboken). 2017 Dec;300(12):2200-2207. doi: 10.1002/ar.23687. Epub 2017 Sep 26. PMID 28921917
- [Background] Gu G, Dubauskaite J, Melton DA. Direct evidence for the pancreatic lineage: NGN3+ cells are islet progenitors and are distinct from duct progenitors. Development. 2002 May;129(10):2447-57. doi: 10.1242/dev.129.10.2447. PMID 11973276
- [Result] Wang L, Fan H, Zhou L, Wu Y, Lu H, Luo J. Altered expression of PGC-1alpha and PDX1 and their methylation status are associated with fetal glucose metabolism in gestational diabetes mellitus. Biochem Biophys Res Commun. 2018 Jun 18;501(1):300-306. doi: 10.1016/j.bbrc.2018.05.010. Epub 2018 May 7. PMID 29730292
- [Result] Plows JF, Stanley JL, Baker PN, Reynolds CM, Vickers MH. The Pathophysiology of Gestational Diabetes Mellitus. Int J Mol Sci. 2018 Oct 26;19(11):3342. doi: 10.3390/ijms19113342. PMID 30373146